CLINICAL TRIAL: NCT00850850
Title: The Use of Physostigmine in Elderly Patients in the Postoperative Recovery-phase After General Anesthesia
Brief Title: Physostigmine After General Anesthesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Frank Pott, ICU
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2006-002497-22
Record Dates: First submitted 2009-02-24; First posted 2009-02-25 (Estimated); Last update posted 2010-05-27 (Estimated); Status verified 2010-05

CONDITIONS: Postoperative Nausea and Vomiting; Anesthesia Recovery Period
Keywords: PACU; Physostigmine; Recovery; Postanesthesia Nursing; Wakefulness; General anesthesia; General Anesthetics; Postoperative Period
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Physostigmine; Sodium Chloride

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Physostigmine (Active Comparator): Patients who have difficulties in awakening from the general anaesthesia and do not suffer from excess nausea or vomiting will be randomised to receive 1 mg of physostigmine.
  Interventions: Drug: physostigmine
- NaCl (Placebo Comparator): Patients who have difficulties in awakening from the general anaesthesia and do not suffer from excess nausea or vomiting will be randomised to receive 1 ml of isotonic sodium chloride solution (placebo).
  Interventions: Drug: Isotonic sodium chloride solution

INTERVENTIONS:
Drug: physostigmine — 1 mg of physostigmine time 0 min. If the condition persisted after 15 min. the same amount of active drug would be administered once again.
  Other Names: Fysostigmin; Methylcarbamate; Erserine; Eserolein
  Arms: Physostigmine
Drug: Isotonic sodium chloride solution — Patients who have difficulties in awakening from the general anaesthesia and do not suffer from excess nausea or vomiting will be randomised to receive 1 ml of isotonic sodium chloride solution (placebo) time 0 min. If the condition persisted after 15 min. the same amount of non-active drug would be administered once again.
  Other Names: NaCl
  Arms: NaCl

SUMMARY:
Recovery after general anaesthesia is often prolonged in the elderly. This group is particularly exposed to post-operative confusion. This has negative personal consequences as well as consequences for the postoperative care for these patients.

The hypothesis is that physostigmine will decrease the amount of time in the post-anaesthesia care unit (PACU ), the postoperative amount of pain and shivering and finally post-operative confusion.

DETAILED DESCRIPTION:
The researchers wish to investigate the use of physostigmine in the elderly patients (age > 60 yrs, ASA I-III) in the postoperative recovery-phase after general anesthesia.

Apart from the beneficial effects for the patient, the lessened amount of time in the PACU will release caregiving resources and thereby increase the efficacy of the PACU.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for surgical acute or elective operation
* General anesthesia.
* ASA physical status I-III
* Age > 60 years

Exclusion Criteria:

* Asthma and chronic pulmonary diseases
* Glaucoma
* Diabetics
* Any history of neurological and psychiatric disorder
* Parkinson's disease
* Disorders of the gastrointestinal and urogenital tracts

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-12; Primary Completion 2011-03 (Estimated); Study Completion 2011-05 (Estimated)

PRIMARY OUTCOMES:
The readiness to be released from the PACU (assessed by the normal guidelines) It should be noted that for safety reasons the patients remained in the PACU for at least 60 minutes | 60 minutes

SECONDARY OUTCOMES:
Pain, shivering and nausea will also be registered on the standardized form as well as a multiple of physiological measurements. A follow-up will be performed after 12 hours from release from the PACU | 6 hours

CONTACTS AND LOCATIONS:
Overall Officials: Frank Pott, MD, Study Director — Bispebjerg Hospital
Locations (1):
- Bispebjerg Hospital, Copenhagen, Copenhagen NV, Denmark